CLINICAL TRIAL: NCT05956470
Title: A Comprehensive Meditation and Breath Program (SKY) as an Adjunct Tool to Increase Resilience and Wellness in Frontline Healthcare Workers - A Randomized Pilot Study
Brief Title: A Comprehensive Wellness Program (SKY) to Mitigate Physician Burnout
Acronym: SKY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Koc University Hospital, Istanbul, Turkey (Unknown); Ataturk Chest Diseases Education and Research Hospital, Ankara, Turkey (Unknown); Izmir Biomedicine and Genome Center (Other Government)
Responsible Party: Principal Investigator, Fahri Saatcioglu, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: iBG-2021-015
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety; Stress; Insomnia; Optimism; Interpersonal Disengagement; Professional Fulfillment; Work Exhaustion; Self-reported Medical Errors; Physician Burnout
Keywords: physician burnout; medical doctor; burnout; stress; depression; wellness; meditation; breathing exercise
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Burnout, Psychological | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The people analysing the results/data were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKY intervention group (Experimental): Meditation and breath program: includes gentle stretches (office yoga' in a sitting position) and three different types of specific breathing exercises. 3x1,5 hours. Daily practice thereafter for about 30 minutes for 8 weeks. In addition, there are weekly one-hour sessions for group practice and discussion.
  Interventions: Behavioral: Meditation and breathing program : Sudarshan Kriya Yoga (SKY)
- Control group (Active Comparator): Group discussion-based viewing of online educational videos that demonstrate ways to mitigate psychological distress, including the use of cognitive coping techniques. 3x1,5 hours. It includes weekly online meetings with group discussions, experience sharing, and watching brief videos on the key elements of the program for 8 weeks.
  Interventions: Behavioral: Stress management education

INTERVENTIONS:
Behavioral: Meditation and breathing program : Sudarshan Kriya Yoga (SKY) — The SKY sessions (3x1,5 h on consecutive days) included online instruction in gentle stretches ('office yoga' in a sitting position), specific breathing exercises and meditation, and discussion of cognitive/behavioral coping skills. After the 3-day program, participants asked to practice the techniques once a day for about 30 min. In addition, there were weekly group exercise sessions of 1 hour where all participants were asked to join.
  Arms: SKY intervention group
Behavioral: Stress management education — This control intervention included viewing of educational videos on stress management and group discussions, where the sessions were equal in length to the SKY intervention. There were also weekly follow-up sessions as in the SKY group where the educational points were reviewed and experiences of the subjects during the previous week was discussed.
  Arms: Control group

SUMMARY:
The primary objective of the study was to determine whether the yoga-based breathing and meditation program SKY could improve wellness indicators in currently practicing physicians. The hypothesis of this study is that SKY is effective in reducing anxiety and depression, increasing subjective optimism, and reducing physician burnout in healthy, actively practicing physicians.

DETAILED DESCRIPTION:
Physicians are exposed to high stress and strain that results in burnout, affecting not only them, their families, patients, but the whole healthcare system. Thus there is an urgent need to develop methods to increase resiliency of physicians. A comprehensive yoga breathing and meditation-based online program (Sudarshan Kriya Yoga, or SKY) is a potential approach to mitigate physician burnout. This is a randomized clinical trial assessing the potential efficacy of SKY compared to a stress management education (SME) training as control, conducted online. Both groups received training for three consecutive days, 1,5 hours per day, through group video conference. Active physicians participated in the study from November 2021 to March 2022. Of the 280 physicians who showed interest and prescreened, 238 were eligible and randomized to receive either the SKY or the control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Actively working physicians without any chronic disease with documented interest in being part of a study to evaluate breath/meditation-derived exercises and a willingness to do some form of relaxation exercises every day for 8 weeks.

Exclusion Criteria:

* Presence of psychiatric illness or other major illnesses, such as bipolar disorder, post-traumatic stress disorder (PTSD), schizophrenia or schizoaffective disorder, uncontrolled hypertension, lung disease, liver disease, cancer, or heart disease; maintaining a regular mind-body program practice such as meditation, yoga, and breathing techniques.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depression, Anxiety, and Stress scale immediately after the intervention and at 8 weeks | At baseline, right after the 3-day intervention, and at 8 weeks post-intervention
  Scores assessed by the Depression, Anxiety, and Stress Scale 42 (DASS-42).
Change from baseline in Professional Satisfaction index post-intervention and at 8 weeks | At baseline, right after the 3-day intervention, and at 8 weeks post-intervention
  Scores assessed by the Professional Satisfaction Index (PFI).
Change from baseline in optimism post-intervention and at 8 weeks | At baseline, right after the 3-day intervention, and at 8 weeks post-intervention
  Optimism scores assessed by the Life Orientation Test (Revised) (LOT-R) and the
Change from baseline in Insomnia post-intervention and at 8 weeks | At baseline, right after the 3-day intervention, and at 8 weeks post-intervention
  Insomnia scores assesed by the Regensburg Insomnia Scale (RIS).

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Biomedicine and Genome Center, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saatcioglu F, Cirit B, Koprucu Suzer G. The Promise of Well-Being Interventions to Mitigate Physician Burnout During the COVID-19 Pandemic and Beyond. JCO Oncol Pract. 2022 Dec;18(12):808-814. doi: 10.1200/OP.22.00108. Epub 2022 Sep 26. PMID 36162039
- [Background] Hlubocky FJ, Symington BE, McFarland DC, Gallagher CM, Dragnev KH, Burke JM, Lee RT, El-Jawahri A, Popp B, Rosenberg AR, Thompson MA, Dizon DS, Srivastava P, Patel MI, Kamal AH, Daugherty CK, Back AL, Dokucu ME, Shanafelt TD. Impact of the COVID-19 Pandemic on Oncologist Burnout, Emotional Well-Being, and Moral Distress: Considerations for the Cancer Organization's Response for Readiness, Mitigation, and Resilience. JCO Oncol Pract. 2021 Jul;17(7):365-374. doi: 10.1200/OP.20.00937. Epub 2021 Feb 8. No abstract available. PMID 33555934
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Background] Cronlein T, Langguth B, Popp R, Lukesch H, Pieh C, Hajak G, Geisler P. Regensburg Insomnia Scale (RIS): a new short rating scale for the assessment of psychological symptoms and sleep in insomnia; study design: development and validation of a new short self-rating scale in a sample of 218 patients suffering from insomnia and 94 healthy controls. Health Qual Life Outcomes. 2013 Apr 22;11:65. doi: 10.1186/1477-7525-11-65. PMID 23601161
- [Derived] Korkmaz A, Bernhardsen GP, Cirit B, Koprucu Suzer G, Kayan H, Bicmen H, Tahra M, Suner A, Lehto SM, Sag D, Saatcioglu F. Sudarshan Kriya Yoga Breathing and a Meditation Program for Burnout Among Physicians: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2353978. doi: 10.1001/jamanetworkopen.2023.53978. PMID 38294813